CLINICAL TRIAL: NCT07299929
Title: Multimodal Physiotherapy Intervention for Active Coping With Persistent Musculoskeletal Pain in Primary Care
Brief Title: Multimodal Physiotherapy and Pain Coping in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Victor Ortiz Mallasen, Assistant Professor of Nursing, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-GVA-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Musculoskeletal Pain
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Physiotherapy Intervention (Experimental): Participants will receive a multimodal physiotherapy intervention designed to improve active coping and health-related quality of life in individuals with persistent musculoskeletal pain. The program combines pain neuroscience education sessions with guided therapeutic exercise, delivered by physiotherapists in Primary Care settings. The intervention will be conducted in group sessions over several weeks and will include education on pain mechanisms, movement retraining, and individualized exercise progression.
  Interventions: Behavioral: Multimodal Physiotherapy Program Based on Pain Neuroscience Education and Therapeutic Exercise

INTERVENTIONS:
Behavioral: Multimodal Physiotherapy Program Based on Pain Neuroscience Education and Therapeutic Exercise — The intervention consists of a multimodal physiotherapy program designed to promote active coping and improve health-related quality of life in patients with persistent musculoskeletal pain. It includes educational sessions on pain neuroscience aimed at reconceptualizing pain and reducing maladaptive beliefs, combined with supervised therapeutic exercise focused on mobility, strength, and functional recovery. The program will be delivered in small group sessions by trained physiotherapists in Primary Care settings over several weeks. Participants will be encouraged to progressively integrate the exercises and concepts into their daily activities to foster self-management and long-term adherence.

SUMMARY:
This quasi-experimental, multicenter study aims to evaluate the effectiveness of a multimodal physiotherapy intervention-based on pain neuroscience education and therapeutic exercise-on health-related quality of life in patients with persistent musculoskeletal pain treated in Primary Care.

The study will be conducted in four Primary Care physiotherapy units in the Valencian Community (Spain). A total of at least 68 participants aged 18 to 70 years with nonspecific persistent musculoskeletal pain lasting at least six months will be recruited.

The intervention will consist of a structured multimodal physiotherapy program including educational sessions on pain neuroscience and guided therapeutic exercise. The main outcome will be health-related quality of life, assessed using the SF-36 Health Survey. Secondary outcomes will include pain catastrophizing (Pain Catastrophizing Scale), kinesiophobia (Tampa Scale for Kinesiophobia), and central sensitization (Central Sensitization Inventory), among others.

Data will be collected using the REDCap electronic platform at three time points: baseline (pre-intervention), immediately after the intervention, and six months post-intervention. Statistical analysis will include descriptive statistics, bivariate analyses, and paired comparisons to assess changes over time.

The study seeks to generate evidence on the feasibility and potential effectiveness of implementing a multimodal physiotherapy intervention for active coping with chronic musculoskeletal pain in the context of Primary Care.

ELIGIBILITY:
Inclusion Criteria:

- Persistent nonspecific musculoskeletal pain lasting at least 6 months

Exclusion Criteria:

* Oncologic pain.
* Spinal fracture or surgical intervention within the 12 months prior to the intervention.
* Cognitive impairment that prevents comprehension of the intervention content (in case of doubt, the Mini-Mental State Examination will be administered, requiring a minimum score of 25).
* Physical performance deficit that prevents execution of the intervention (minimum requirement: completion of the Timed Up and Go test within the normal time of 10 seconds).
* Pregnancy.
* Cauda equina syndrome.
* Presence of urinary and/or fecal incontinence.
* Severe psychiatric disorders.
* Autoimmune diseases.
* Associated medical conditions that preclude participation in a physical exercise program (e.g., myopathies, neurological diseases with significant functional impairment).
* Patients undergoing alternative therapies.
* Patients with an implanted neurostimulator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life Measured With the 36-Item Short Form Health Survey (SF-36) | Baseline (before the intervention), immediately after the intervention, and 6 months after the intervention.
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). The instrument provides eight domain scores and a total score, each ranging from 0 to 100. Higher scores indicate better perceived health-related quality of life.

SECONDARY OUTCOMES:
Pain Catastrophizing Measured With the Pain Catastrophizing Scale (PCS) | Baseline (before the intervention), immediately after the intervention, and 6 months after the intervention.
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), a 13-item questionnaire evaluating rumination, magnification, and helplessness related to pain. Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.
Kinesiophobia Assessed Using the Tampa Scale for Kinesiophobia (TSK-11 or TSK-17) | Baseline (before the intervention), immediately after the intervention, and 6 months after the intervention.
  Kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK), a validated questionnaire measuring fear of movement and reinjury. Higher scores indicate greater kinesiophobia.
Central Sensitization Assessed With the Central Sensitization Inventory (CSI) | Baseline (before the intervention), immediately after the intervention, and 6 months after the intervention.
  Central sensitization will be assessed using the Central Sensitization Inventory (CSI), a 25-item questionnaire evaluating symptoms associated with central sensitivity syndromes. Scores range from 0 to 100, with higher scores indicating greater central sensitization.
Pain Intensity Measured Using the Numerical Rating Scale (NRS 0-10) | Baseline (before the intervention), immediately after the intervention, and 6 months after the intervention.
  Pain intensity will be measured using the 11-point Numerical Rating Scale (NRS), where participants rate their average pain during the previous week from 0 ("no pain") to 10 ("worst imaginable pain"). Higher scores indicate greater pain intensity.
Treatment Adherence Assessed With a Session Attendance Log | During the intervention period
  Treatment adherence will be assessed by recording the number of intervention sessions attended by each participant, expressed as the percentage of sessions completed relative to the total scheduled.
Patient Satisfaction Measured With a Likert-Type Satisfaction Questionnaire | Immediately after the intervention.
  Patient satisfaction with the intervention will be assessed using a Likert-type questionnaire (e.g., 0-10 scale or 5-point scale). Higher scores indicate greater satisfaction.

IPD SHARING:
Plan to Share IPD: No